CLINICAL TRIAL: NCT03439371
Title: A Phase II, Multicenter, Open Label Study Evaluating the Efficacy and the Tolerance of Micro-transplantation in Elderly Patients With Acute Myeloid Leukemia (MTSA)
Brief Title: Micro-transplantation in Elderly Patients With Acute Myeloid Leukemia
Acronym: MTSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1201; 2017-A03572-51 (Other: ANSM)
Record Dates: First submitted 2018-02-05; First posted 2018-02-20 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Micro-transplantation; Elderly; Graft-versus-leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HLA-mismatched micro-transplantation (Experimental): HLA-mismatched micro-transplantation
  Interventions: Other: HLA-mismatched micro-transplantation after induction chemotherapy

INTERVENTIONS:
Other: HLA-mismatched micro-transplantation after induction chemotherapy — HLA-mismatched micro-transplantation after induction chemotherapy

SUMMARY:
This study aims at evaluating the safety and the tolerance of the micro-transplantation in elderly patients with acute myeloid leukemia who are ineligible to conventional allogeneic transplantation.

DETAILED DESCRIPTION:
Acute Myeloid Leukemia (AML) is an aggressive hematological malignancy with a median age at diagnosis of 65 years. Outcomes of AML in elderly population remain unsatisfactory with low rates of complete remission, poor disease-free and overall survival. Therapeutic management of older patients with AML deals with patient-related features (i.e. comorbid conditions and performance status) as well as disease-related prognostic factors (i.e. cytogenetics and molecular genetics). Even if allogeneic hematopoietic-cell transplantation provides the strongest antineoplasic effect, this treatment option remains limited for older patients owing to toxicities, the development of significant graft-versus-host disease (GVHD) and logistics of donor availability. More recently, micro-transplantation has emerged as an alternative strategy based on the infusion of mobilized HLA-mismatched related donor cells after induction chemotherapy, thus exerting a graft-versus-leukemia effect without substantial donor engraftment and GVHD. Therefore, there is much of interest in investigating the efficacy and the safety of this method for older patients with AML who are not candidates for allogeneic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated to a social security regimen or beneficiary of the same
* Signed written informed consent form
* Patient, ≥ 60 years-old - < 75 years-old, with established diagnosis of de novo or secondary AML with intermediate-risk or adverse-risk cytogenetic profile, or with established myelodysplasic syndromes (RAEB), in pathologically confirmed complete remission following anti-leukemic induction therapy (<5% blasts)
* Contra-indication to conditioning regimen in conventional allogeneic transplantation

Exclusion Criteria:

* Patient with established diagnosis of acute myeloid leukemia with standard-risk cytogenetic profile
* Promyelocytic leukemia t(15;17)
* CBF-AML t(8;21) or inv(16)
* Normal karyotype with a favorable molecular profile: NPM1+ and FLT3-; NPM1+, FLT3- and double mutation CEBPα or chronic myeloid leukemia in blastic phase
* Patient under guardianship or deprived of his liberty or any condition that may affect the patient's ability to understand and sign the informed consent
* Refusing participation

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of overall survival | 2 years
  Rate of overall survival will be reported.

SECONDARY OUTCOMES:
Hematopoietic recovery | 3 months
  Number of platelets will be reported.
Hematopoietic recovery | 3 months
  Number of neutrophils will be reported.
Hematopoietic recovery | 3 months
  Percentage of leukaemic blasts will be reported.
Rate of complete remission | 2 years
  Rate of complete remission :
GVHD (graft versus host disease) | 2 years
  Presence of graft versus host disease will be reported.
Median overall survival | 2 years
  Median overall survival will be calculated.
Median progression-free survival | 2 years
  Median progression-free survival will be calculated.
Microchimerism | 3 months
  Presence of microchimerism will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Cornillon, MD, Principal Investigator — CHU de Saint-Etienne
Locations (7):
- France (7):
  - CHU Estaing, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - CHRU de Lille, Lille
  - Centre Hospitalier Lyon Sud, Lyon
  - Centre Hospitalier Universitaire de Nancy, Nancy
  - Hôpital de la Pitié-Salpêtrière, Paris
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No